CLINICAL TRIAL: NCT06148116
Title: Attitudes and Knowledge of Dialysis Patients Towards Kidney Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Paulina Kurleto, PhD, Andrzej Frycz Modrzewski Krakow University
Other Study IDs: KAAFMWLNZ/34/0/2023
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Poland, approximately 4.2 million people suffer from chronic kidney disease [1]. In December 2022, a total of 20,198 patients were dialyzed in the country, of which 96% by hemodialysis (HD) and 4% by peritoneal dialysis (DO). In 2022, kidney transplantation was performed in 2.6% of patients dialyzed using the HD method and in 15.4% of patients dialyzed using the DO method [2]. According to the data of the Organizational and Coordination Center for Transplantation "Poltransplant", in 2022 on the national waiting list 1,119 people were registered for kidney transplantation. The average age of those waiting was 49 years [3]. In Poland, according to data from 2022, the average waiting time for transplantation in the case of the first transplant from the moment of registration on the waiting list was 387 days, and 1,106 days from the start of dialysis. Data show that only 5.5% of patients undergoing renal replacement therapy are on the waiting list [3].

Therefore, a study was designed to examine the knowledge and attitudes towards kidney transplantation among dialysis patients. The study will include a representative group of dialysis patients from all voivodeships and aims to identify positive and negative aspects related to patients' attitudes towards kidney transplantation.

The scientific value of the study is worth emphasizing, because so far in Poland no research has been conducted on the knowledge and attitudes towards kidney transplantation among dialysis patients in all voivodeships in the country. The study will identify the level of knowledge and attitudes of dialysis patients towards transplantation. The results of this study may contribute to the development and implementation of new educational and information programs that may increase the level of knowledge and influence attitudes towards transplantation, which may largely contribute to the increase in transplantation among people with chronic kidney disease.

References:

1. Gellert R, Durlik M, Małgorzewicz S. Raport 2019. Ogólnopolskie Badanie Pacjentów Nefrologicznych. Forum Nefrologiczne. 2020;13(3):149-63.
2. Dębska-Ślizień A, Rutkowski B, Rutkowski P et al. (2022). Aktualny stan leczenia nerkozastępczego w Polsce-2022. Nefrol Dializoter Pol, 26: 21-38.
3. Centrum Organizacyjno- Koordynacyjne do spraw transplantacji-Poltransplant. Biuletyn Informacyjny 2023. https://files.poltransplant.org.pl/Biuletyn_2023_www.pdf Accessed 13 November 2023.

ELIGIBILITY:
Inclusion Criteria:

(1) patients on dialysis for at least 3 months; (2) patients who have no medical contraindications to kidney transplantation and patients who are temporarily suspended from KLO; (3) voluntary consent to participate in the study; (4) communicative knowledge of Polish

Exclusion Criteria:

(1) inability to make an informed and independent decision; (2) patients with absolute medical contraindications to kidney transplantation, i.e. recently diagnosed or disseminated cancer, persistent untreated infection, severe irreversible systemic disease, expected short life span, lack of cooperation (alcohol and drug addiction, mental illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People undergoing dialysis in all voivodeships in Poland
  .
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Attitudes and Knowledge of Dialysis Patients Towards Kidney Transplantation | 16 months
  Attitudes and Knowledge will be measured using a 51-item self-report questionnaire with single and multi-choice questions.
Intensity of pain and attitudes towards kidney transplantation. | 16 months
  To investigate the relationship between the intensity of pain in dialysis patients and their attitudes towards kidney transplantation.
  Standardized tool will be the Numeric Rating Scale (NRS). Pain intensity will be assessed using the NRS, where 0 meant no pain and 10 maximum pain. Numeric scores of 1-3, 4-6, and 7-10 corresponded to mild, moderate and severe pain
Anxiety and Depression | 16 months
  To investigate the relationship between the level of anxiety and depression of dialysis patients and their attitudes towards kidney transplantation.
  Emotional state will be evaluated using HADS [21, 22], which was validated for Polish conditions. It consists of 7 items grouped in sub-scales: anxiety and depression. The answers describe the patient's well-being over the last week and are coded on a scale of 0-3 points. The total score amounts to 0-21 points (0-7 points = norm, 8-10 = borderline, ≥11 points = clinical levels of symptoms).
Acceptance of the disease | 16 months
  To measure it, the Acceptance of Illness Scale (AIS), by Felton, Revenson and Hinrichsen, in the Polish adaptation by Juczyński was used [4]. It consists of 8 questions describing the consequences of poor health. The questions concerned the limitations imposed by the disease, lack of self-sufficiency, feeling of dependence on others and reduced self-esteem. Questions contained a five-point scale, and the person described their current health condition by marking the number: 1 - I strongly agree, 2 - I agree, 3 - I don't know, 4 - I disagree, 5 - I strongly disagree. Strong consent meant poor adaptation to the disease, while lack of consent meant acceptance of the disease. The degree of acceptance of the current health condition was the sum of all points, ranging from 8 to 40 points. Three point ranges were created to determine the degree of acceptance, where the number of points: 8-18 meant lack of acceptance of the disease, 19-29 - average acceptance, 30-40 - good acceptance.
Patient Request Form | 16 months
  To investigate the relationship between patient expectations and their attitudes towards kidney transplantation. Patient expectations will be measured using the Patient Request Form - the scale consists of 18 statements regarding expectations towards the doctor/medical staff related to explaining the disease, seeking support and obtaining information about tests and treatment. The theoretical range of the scale is from 0 to 12 points. The higher the score, the greater the patient's expectations for specific help.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Kurleto, PhD, Study Director — Andrzej Frycz Modrzewski Krakow University
Locations (1):
- Andrzej Frycz Modrzewski Krakow University, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kurleto P, Tomaszek L, Milaniak I, Debska G, Turkanik E, Siekierska B, Danielewicz R, Debska-Slizien A, Pietrzyk JA. Factors associated with the willingness to become a kidney transplant recipient horizontal line the results from a national cross sectional study. BMC Nephrol. 2025 Oct 16;26(1):571. doi: 10.1186/s12882-025-04516-2. PMID 41102657